CLINICAL TRIAL: NCT03815630
Title: Clinical Study on the Safety and Efficacy of Pd-1 Combined With Dc-cik in the Treatment of Solid Tumors
Brief Title: A Study of PD1 Combined With Dc-cik in the Treatment of Solid Tumors
Acronym: DC-CIK
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Yunnan Province/First People's Hospital of Yunan Provinve New Kunhua Hospital (Unknown); Henan Provincial People's Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PD-1/DC CIK-YNYY-01
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — alpha-Synuclein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 and dc-cik treatment group (Experimental)
  Interventions: Drug: pd-1 and dc-cik cells

INTERVENTIONS:
Drug: pd-1 and dc-cik cells — Total dose of 10ml Keytruda will be administered at day0, 60million DC cells and 1.5 billion CIK at day1, 1.5 billion CIK cells at day2, 1.5 billion CIK cells at day3 .

SUMMARY:
This is a single center、single arm、open-label, to investigate the safety and efficacy of PD-1 and DC-CIK with anti-solid tumor

ELIGIBILITY:
Inclusion Criteria:

1. Previously receiving ≥ first-line regimen chemotherapy;
2. Age over 3 years old and less than 14 years old;
3. The expected survival period is more than 3 months;
4. ECOG≤2;
5. Vital organ function is satisfied: cardiac ultrasound indicates cardiac ejection fraction ≥ 50%, no obvious abnormality in ECG; blood oxygen saturation ≥ 90%; creatinine clearance calculated by Cockcroft-Gault formula ≥ 40ml/min; ALT and AST ≤ 3 times the normal range, total bilirubin ≤ 2.0 mg / dl;
6. Blood routine: Hgb≥80g/L, ANC≥1×109/L, PLT≥50×109/L;
7. There are measurable target lesions.

Exclusion Criteria:

1. Liver and kidney function:

   * Total bilirubin > 2 x ULN (Gilbert syndrome > 3 x ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 3 × ULN
   * Serum creatinine clearance >60mL/min
2. Serological examination:

   * Absolute neutrophil count (ANC) <0.75x109/L
   * Platelet count (PLT) <50x109/L
3. Active hepatitis B (HBV-DNA > 1000 copies / ml), hepatitis C, or uncontrolled infection;
4. The number of days of chemotherapy medication and the administration of hormones below 5mg is ≤3, and the number of days of withdrawal of hormones greater than 5mg is ≤5;
5. Active CNS disease (tumor cells in CSF);
6. Intracranial hypertension or unconsciousness; respiratory failure; diffuse vascular internal coagulation;
7. creatinine > 1.5 times the upper limit of normal or ALT / AST > 3 times the upper limit of normal or bilirubin > 2 times the upper limit of normal;
8. The New York Heart Association (NYHA) is classified as Level III or higher;
9. Uncontrolled diabetes;
10. With other uncontrolled diseases, the investigator believes that it is not suitable for joining;
11. Any situation that the investigator believes may increase the risk of the subject or interfere with the test results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
occurrence of treatment related adverse events | 1 year
  occurrence of treatment related adverse events that are possible, likely. Or definitely related to study treatment.

IPD SHARING:
Plan to Share IPD: No